CLINICAL TRIAL: NCT03082209
Title: An Open-Label, Phase 1, First-In-Human Study of TRAIL Receptor Agonist ABBV-621 in Subjects With Previously-Treated Solid Tumors and Hematologic Malignancies
Brief Title: A Study of the Safety and Tolerability of ABBV-621 in Participants With Previously-Treated Solid Tumors and Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-913; 2016-003887-37 (EudraCT Number)
Record Dates: First submitted 2017-03-14; First posted 2017-03-17 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumors; Cancer; Hematologic Malignancies
Keywords: Solid Tumors; Hematologic Malignancies; Cancer; non-Hodgkin lymphoma; acute myeloid leukemia (AML); colorectal cancer (CRC); Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Colorectal Neoplasms; Lymphoma, Large B-Cell, Diffuse | interventions — venetoclax; Bevacizumab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Chemotherapy combination: ABBV-621 + FOLFIRI + Bevacizumab (Experimental): Participants with KRAS-mutant CRC are administered with ABBV-621 in combination with bevacizumab plus FOLFIRI
  Interventions: Drug: ABBV-621; Drug: Bevacizumab; Drug: FOLFIRI
- Chemotherapy combination: ABBV-621+FOLFIRI (Experimental): Participants with RAS-mutant CRC who have received one prior line of therapy will be administered ABBV-621 in combination FOLFIRI.
  Interventions: Drug: ABBV-621; Drug: FOLFIRI
- Dose Optimization: ABBV-621 + Venetoclax for AML (Experimental): Additional participants with AML will be enrolled and will be treated with a combination of ABBV-621 and venetoclax.
  Interventions: Drug: ABBV-621; Drug: Venetoclax
- Dose Optimization: ABBV-621 Monotherapy for AML (Experimental): Participants with Acute Myeloid Leukemia (AML) will be treated with ABBV-621 monotherapy.
  Interventions: Drug: ABBV-621
- Dose Optimization: ABBV-621 + Venetoclax for DLBCL (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) will be treated with a combination of ABBV-621 and venetoclax.
  Interventions: Drug: ABBV-621; Drug: Venetoclax
- Dose Optimization for Pancreatic Cancer (Experimental): Participants with pancreatic cancer will be treated with single-agent ABBV-621 to enable selection of the recommended Phase 2 dose (RP2D).
  Interventions: Drug: ABBV-621
- Dose Optimization for KRAS-mutant CRC (Experimental): Participants with colorectal cancer (CRC) will be treated with single-agent ABBV-621 to enable selection of the RP2D.
  Interventions: Drug: ABBV-621
- Dose Escalation (Experimental): ABBV-621 via intravenous administration at escalating dose levels in participants with solid tumors including Non-Hodgkin Lymphoma (NHL).
  Interventions: Drug: ABBV-621

INTERVENTIONS:
Drug: ABBV-621 — Intravenous (IV)
Drug: Venetoclax — tablet, oral
  Other Names: ABT-199; GDC-0199
  Arms: Dose Optimization: ABBV-621 + Venetoclax for AML; Dose Optimization: ABBV-621 + Venetoclax for DLBCL
Drug: Bevacizumab — IV infusion
  Arms: Chemotherapy combination: ABBV-621 + FOLFIRI + Bevacizumab
Drug: FOLFIRI — IV infusion
  Arms: Chemotherapy combination: ABBV-621 + FOLFIRI + Bevacizumab; Chemotherapy combination: ABBV-621+FOLFIRI

SUMMARY:
This is an open-label, Phase I, dose-escalation study to determine the maximum tolerated dose (MTD) and/or recommended phase two dose (RPTD), and evaluate the safety, efficacy, and pharmacokinetic (PK) profile of ABBV-621 for participants with previously-treated solid tumors or hematologic malignancies.

Only chemotherapy combination (ABBV-621 + FOLFIRI) enrolling participants with RAS-mutant CRC who have received one prior line of therapy is open for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of a solid tumor (except primary brain tumors), acute myeloid leukemia (AML), or non-Hodgkin lymphoma (NHL); NHL may be of any subtype for Dose Escalation but is limited to diffuse large B-cell lymphoma (DLBCL) for those enrolled to the cohort evaluating the combination of ABBV-621 and venetoclax. Participants in the Dose Optimization solid tumor cohorts must have either colorectal cancer with documented KRAS mutations (as determined by local testing), or pancreatic cancer (irrespective of mutational status). Participants in the chemotherapy combination cohorts must have metastatic or advanced unresectable colorectal cancer with documented RAS mutations (as determined by local testing).
* Participant in dose escalation or dose optimization cohort must have received at least one prior systemic therapy, and must have relapsed or progressed after, or failed to respond to any/all available effective therapy or therapies.
* Participant in chemotherapy cohorts with CRC must have progressed after or failed to respond to initial systemic therapy.
* Must have measurable disease (by Response Evaluation Criteria In Solid Tumors [RECIST] 1.1 for those with solid tumors; by Lugano classification for those with NHL), except those with AML, who must have histologically confirmed relapsed or refractory disease.
* Must agree to provide the following samples for biomarker analysis:

  * All participants: archived tumor tissue (if available).
  * Participants in Dose Optimization (excluding AML): pre- and on-treatment fresh tissue biopsies. (Note: fresh tissue biopsies will be optional for participants with solid tumor or NHL in Dose Escalation and will be collected only if consent is provided)
  * All participants with AML: pre- and on-treatment bone marrow aspirates (BMA)
  * Participants in chemotherapy combination cohorts: participants must provide a fresh biopsy if an archival biopsy is not available
* Participant in chemotherapy cohorts with CRC must have confirmed RAS mutation
* Must have an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 - 2. Participants in chemotherapy combination cohorts must have ECOG Performance Score of 0 - 1.
* Must have adequate hematologic, renal and hepatic function.

Exclusion Criteria:

* Participants with history of brain metastases who have not shown clinical and radiographic stable disease for at least 28 days after definitive therapy. In addition, any AML participant identified through cerebrospinal fluid (CSF) analysis, as having active central nervous system (CNS) disease, will be excluded.
* Presence of primary hepatobiliary malignancy, including cholangiocarcinoma or hepatocellular carcinoma, gallbladder carcinoma, cancer of ampulla of Vater.
* Receipt of any systemic anti-cancer agent, including investigational anti-cancer products, within 21 days prior to study drug administration or 3 half-lives, whichever is longer.
* Participant with a history of cirrhosis or other indication of significant possible hepatic dysfunction. Note: Those with non-alcoholic steatohepatitis (NASH) should be discussed with the AbbVie TA MD before enrollment.
* Participant with a positive diagnosis of hepatitis A, B, or C.
* Dose Optimization combination cohorts only: Prior receipt, at any time, of a BCL-2 inhibitor
* Dose Optimization combination cohorts only: Participant has received strong or moderate CYP3A inhibitors or inducers within 7 days prior to the initiation of study treatment.
* Dose Optimization combination cohorts only: Participant has malabsorption syndrome or other condition that precludes enteral route of administration.
* Dose Optimization combination cohorts only: Participant has promyelocytic leukemia (M3).
* CRC chemotherapy cohort only: Participant with minor surgical procedures, such as fine needle aspirations or core biopsies, within 7 days prior to first dose of study drug are excluded.
* Participants in CRC chemotherapy combination cohort only: cardiomyopathy, coronary/peripheral artery bypass graft, aneurysm or aneurysm repair, angioplasty, pulmonary hypertension, cerebrovascular accident or transient ischemic attack, within 1 year of first dose of study drug.
* Chemotherapy combination CRC participants only: Prior receipt of an irinotecan-based chemotherapy.
* Chemotherapy combination CRC participants only: Disease progression within 3-months of initiating first-line therapy.
* Chemotherapy combination CRC participants only: history of Gilbert's syndrome or UG1T1A1 genotypes.
* Chemotherapy combination with bevacizumab participants only: clinically significant conditions that may place the participant at higher risk with anti-angiogenic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) for ABBV-621 | Up to 21 days
  The MTD and/or RP2D of ABBV-621 will be determined during the dose escalation phase of the study of ABBV-621
Area under the serum/plasma concentration time curve (AUC) of ABBV-621 | Up to 64 days
  Area under the serum/plasma concentration time curve (AUC) of ABBV-621.
Area under the serum/plasma concentration time curve (AUC) of Venetoclax | Up to 64 days
  Area under the serum/plasma concentration time curve (AUC) of venetoclax.
Maximum observed serum concentration (Cmax) of ABBV-621 | Up to 64 days
  Maximum observed serum concentration (Cmax) of ABBV-621.
Maximum observed serum concentration (Cmax) of Venetoclax | Up to 64 days
  Maximum observed serum concentration (Cmax) of venetoclax.
Time to Cmax (Tmax) of ABBV-621 | Up to 64 days
  Time to Cmax (Tmax) of ABBV-621.
Time to Cmax (Tmax) of Venetoclax | Up to 64 days
  Time to Cmax (Tmax) of ventoclax.
Terminal phase elimination rate constant (β) for ABBV-621 | Up to 64 days
  Terminal phase elimination rate constant (β) for ABBV-621.
Terminal phase elimination rate constant (β) for Venetoclax | Up to 64 days
  Terminal phase elimination rate constant (β) for venetoclax.
Terminal Phase Elimination Half-life (t1/2) of ABBV-621 in Plasma | Up to 64 days
  Terminal phase elimination half-life (t1/2) for ABBV-621.
Terminal Phase Elimination Half-life (t1/2) of Venetoclax in Plasma | Up to 64 days
  Terminal phase elimination half-life (t1/2) for venetoclax.

SECONDARY OUTCOMES:
QTcF Change from Baseline | Up to 64 days
  QT interval measurement corrected by Fridericia's formula (QTcF) mean change from baseline by dose level
Number of Participants with Dose-limiting Toxicities (DLTs) | Up to 42 days after first day of study drug administration or 14 days after bone marrow biopsy showing < 5% blast count (whichever is later)
  Dose limiting toxicities for dose escalation purposes will be determined on events that occur during the first 21-day cycle (with protocol specified exceptions for AML participants).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (19):
- United States (10):
  - Yale University /ID# 158029, New Haven, Connecticut
  - The University of Chicago Medical Center /ID# 158030, Chicago, Illinois
  - Ingalls Memorial Hosp /ID# 171221, Harvey, Illinois
  - Univ Michigan Med Ctr /ID# 207134, Ann Arbor, Michigan
  - Rhode Island Hospital /ID# 171157, Providence, Rhode Island
  - Vanderbilt University Medical Center /ID# 215000, Nashville, Tennessee
  - MD Anderson Cancer Center /ID# 202187, Houston, Texas
  - Millennium Oncology /ID# 214981, Houston, Texas
  - South Texas Accelerated Research Therapeutics /ID# 160574, San Antonio, Texas
  - Medical College of Wisconsin /ID# 171152, Milwaukee, Wisconsin
- Japan (2):
  - National Cancer Center Hospital East /ID# 160596, Kashiwa-shi, Chiba
  - Yamagata University Hospital /ID# 200681, Yamagata, Yamagata
- Netherlands (4):
  - Erasmus Medisch Centrum /ID# 160869, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen /ID# 169748, Groningen
  - Maastricht Universitair Medisch Centrum /ID# 214935, Maastricht
  - Universitair Medisch Centrum Utrecht /ID# 169747, Utrecht
- Spain (3):
  - Hospital Universitario Vall d'Hebron /ID# 170809, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 200106, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 165136, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biesdorf C, Guan X, Siddani SR, Hoffman D, Boehm N, Medeiros BC, Doi T, de Jonge M, Rasco D, Menon RM, Polepally AR. Pharmacokinetics and immunogenicity of eftozanermin alfa in subjects with previously-treated solid tumors or hematologic malignancies: results from a phase 1 first-in-human study. Cancer Chemother Pharmacol. 2024 Apr;93(4):329-339. doi: 10.1007/s00280-023-04613-9. Epub 2023 Nov 30. PMID 38036720
- [Derived] Tahir SK, Calvo E, Carneiro BA, Yuda J, Shreenivas A, Jongen-Lavrencic M, Gort E, Ishizawa K, Morillo D, Biesdorf C, Smith M, Cheng D, Motwani M, Sharon D, Uziel T, Modi DA, Buchanan FG, Morgan-Lappe S, Medeiros BC, Phillips DC. Activity of eftozanermin alfa plus venetoclax in preclinical models and patients with acute myeloid leukemia. Blood. 2023 Apr 27;141(17):2114-2126. doi: 10.1182/blood.2022017333. PMID 36720090
- [Derived] LoRusso P, Ratain MJ, Doi T, Rasco DW, de Jonge MJA, Moreno V, Carneiro BA, Devriese LA, Petrich A, Modi D, Morgan-Lappe S, Nuthalapati S, Motwani M, Dunbar M, Glasgow J, Medeiros BC, Calvo E. Eftozanermin alfa (ABBV-621) monotherapy in patients with previously treated solid tumors: findings of a phase 1, first-in-human study. Invest New Drugs. 2022 Aug;40(4):762-772. doi: 10.1007/s10637-022-01247-1. Epub 2022 Apr 25. PMID 35467243